CLINICAL TRIAL: NCT04020536
Title: Real World Study of Classic Infectious Disease
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); The ninth Hospital of NanChang city (Unknown); Luoyang Central Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); The Fifth Affiliated Hospital Xinjiang Medical University (Unknown); LanZhou University (Other); Huzhou Central Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Fuzhou Municipal Infectious Diseases Hospital (Unknown); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Lanzhou Medical University (Unknown); Linyi People's Hospital (Other); Nantong University (Other); Nanyang Central Hospital (Other); Qilu Hospital of Shandong University (Other); Qianfoshan Hospital (Other); Infectious Hospital of Jining City (Unknown); The Affiliated Hospital of Jining Medical University and Zaozhuang City (Unknown); The First Affiliated Hospital of Shanxi Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Yuncheng Central Hospital (Other); Zibo Central Hospital (Other Government); The Second Affiliated Hospital of Henan Medical University (Unknown); West Hospital of the First Affiliated Hospital of Guangxi University (Unknown); The First Hospital of Jilin University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Second Hospital of Shandong University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Chief of dpartment of infectious disease, Huashan Hospital
Other Study IDs: KY2019-RWS(CID)
Record Dates: First submitted 2019-07-06; First posted 2019-07-16 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Brucelloses; Epidemic Hemorrhagic Fever; Kala-Azar
Keywords: real world study
MeSH Terms: conditions — Brucellosis; Hemorrhagic Fever with Renal Syndrome; Leishmaniasis, Visceral | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- kala-azar group
  Interventions: Drug: Antibiotics
- epidemic hemorrhagic fever group
  Interventions: Drug: Antibiotics
- brucellosis group
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — Local doctors prescribe available antibiotics to the patients according to the guideline and patients' condition

SUMMARY:
This study aimed to collect and analyze clinical specimens of patients with classic infectious diseases in the real world. To investigate the epidemiological distribution of classic infectious diseases (brucellosis, epidemic hemorrhagic fever, kala-azar) and treatment options suitable for China.

DETAILED DESCRIPTION:
Brucellosis is present in humans and animals in nearly 170 countries and regions around the world. In the 1950s and 1960s, brucellosis was seriously prevalent in China. In the 1970s, the epidemic gradually declined. It was basically controlled in the 1980s and early 1990s, but since the mid-1990s, the epidemic has continued to rise rapidly, and brucellosis It has become one of the fastest infectious diseases reporting the rising incidence rate. In 2016, 47,139 cases were reported, with an incidence rate of 3.44/100,000. The provinces with the most reported cases are Xinjiang Uygur Autonomous Region, Inner Mongolia Autonomous Region, Shanxi Province and Heilongjiang Province. However, in the southern non-pastoral areas of Guangdong Province and Guangxi Province, brucellosis outbreaks have occurred in recent years, and the incidence rates in Henan and Fujian provinces have continued to rise.

Hemorrhagic fever with renal syndrome, also known as epidemic hemorrhagic fever, is an infectious disease caused by the Hantavirus. The main clinical features are fever, exudation, hemorrhage, hypotensive shock, and kidney damage. It was once epidemic viral infection in China after viral hepatitis. In the 1980s, the number of cases reported exceeded 100,000. More than 1650,000 patients have been reported in China since 1950, including more than 47,000 deaths, with a total case fatality rate of approximately 2.89%. The number of people in the province accounted for more than 80% of the total number of people in the country. From 2004 to 2015, Shaanxi Province and the three northeastern provinces were the hardest hit areas of national hemorrhagic fever.

There are reports of sporadic leishmaniasis in China, but they are rare and lack corresponding epidemiological data. In 2015, 507 new cases of visceral leishmaniasis were reported, which was a high level in the past 10 years. However, the incidence rate remains at a low level of 0.0372/100,000. In recent years, visceral leishmaniasis is mainly distributed in the northwestern part of China, and there are many cases reported in the southwestern part of the country. The three areas with the highest incidence rate are Xinjiang Uygur Autonomous Region, Gansu Province and Sichuan Province. The cases in non-endemic areas are mainly adults who go to work in popular areas, and mainly male physical workers, while the popular areas are mainly infants and young children.

ELIGIBILITY:
Inclusion Criteria:

Brucellosis： Patients with any of the following confirmed the evidence.

1. sample culture: Brucella;
2. Specific antigen or antibody (IgG or IgM) positive. epidemic hemorrhagic fever：

1 specific antibody positive 2 Hantavirus RNA positive kala-azar：

1. latent infection: rK39 antibody positive
2. patients with the following evidence of kala-azar diagnosis: 1) bone marrow, spleen puncture sample culture: Leishmania; 2) bone marrow, spleen puncture sample smear: Leishmania; 3) clinical symptoms, history of exposure or epidemiology, and positive screening test (rK39 positive)

Exclusion Criteria:

1. Patient history data is incomplete
2. HIV antibody positive and AIDS patients
3. Patients who participated in other clinical trials during the same period.
4. Pregnant, lactating women or women of childbearing age who are ready to conceive.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This research plans to enroll 10000 outpatients or hospitalized patients (≥ 18 years old with the main diagnosis as classic infectious disease).Hospital selection follows a multi-stage sampling strategy.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-05-13 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients With Prevalence Rate of specific infectious diseases(brucellosis, epidemic hemorrhagic fever, and kala-azar） | 1 day

SECONDARY OUTCOMES:
Number of Participants With Successful Treatment of specific antibiotic therapy. | 30 days
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li D, Yuan G, Wang YO, Wang H, Zhang Q, Wang YA, Gu Y, Zhang H, Zhang Y, Song J, Fu Z, Lin K, Qiu C, Zhou Y, Fan M, Zhao Y, Guo J, Jiang N, Ai J, Liu H, Zhang W. Clinical Characteristics, Treatment, and Prognosis of Osteoarticular Brucellosis: A Retrospective Real-World Study in Shenyang, China, 2014-2019. Foodborne Pathog Dis. 2025 Feb;22(2):86-96. doi: 10.1089/fpd.2023.0027. Epub 2024 Apr 12. PMID 38608217